CLINICAL TRIAL: NCT04831346
Title: Effects of Low-Level Laser Therapy Versus Soft Occlusive Splints on Mouth Opening and Surface Electromyography in Temporomandibular Disorders
Brief Title: Effects of Low-Level Laser Therapy on Mouth Opening and Surface Electromyography in Temporomandibular Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tamer Mohamed Shousha, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU2020
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome; Pain, Face
Keywords: Temporomandibular; Dysfunction; VAS; EMG; Laser
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Facial Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment A prospective, parallel-group, randomized clinical trial participants will be randomly assigned to the control group or one of the 2 intervention groups. One group received low level laser therapy (gallium arsenide diode ) while the other received the soft occusive splint. The control group was considered as a wait list for laser treatment aand did not recieve any treatment during the intervention period.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants as well as The assessor, who took the measurements for both the intervention and control groups, was blinded to the subject's group, while the treating therapist was not blinded to the treatment intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low level laser (Experimental): A low-level gallium arsenide diode (Biolase, USA) at a 940 nm wavelength with 0.2 W output power and 2 J energy. The device was calibrated, and the probe was disinfected prior to every treatment.
  The Masseter and Temporalis muscles will be bilaterally assessed with constant pressure to define tenderness.
  LLLT applied perpendicular to each tender point of the intended muscles for 10 seconds with an energy density of 2.5 J/cm2.
  Sessions are scheduled 3 days a week (every other day)
  Interventions: Other: Low level laser
- Occlusive splint therapy (Experimental): A soft occlusal splint (vacuum-formed ) made from a 2-mm-thick elastic rubber sheets will be used.
  Splints were individually designed ( in the out patient clinic of the college of dentistry) for the upper arch of each patient. An alginate imprint of the maxillary arch will be taken to fabricate a master cast of the maxilla.
  A vacuum pressure device was utilized for molding the rubber sheets (13 x 13 cm /2-mm thickness).
  Sheets were removed after it has been appropriately adjusted to the mold in the vacuum former. Edges will be properly trimmed, and the palate part is detached to obtain the end shape.
  Participants are instructed to wear the splint at all times except during mealtimes and oral hygiene.
  Interventions: Device: Soft occlusive splint
- Control (No Intervention): This group will be a wait list group recieving no intervention except for the regular analgesic prescribed by the reffering dentist

INTERVENTIONS:
Other: Low level laser — 940 nm wavelength with 0.2 W output power and 2 J energy applied for 10 seconds with an energy density of 2.5 J/cm2.
  Other Names: A low-level gallium arsenide diode
  Arms: low level laser
Device: Soft occlusive splint — A vacuum-formed soft occlusal splint made from a 2-mm-thick elastic rubber sheets.
  Participants are instructed to always wear the splint except during mealtimes and oral hygiene.
  Arms: Occlusive splint therapy

SUMMARY:
This is a one year followup study that aims to assess the efficacy of low level laser therapy (LLLT) on pain, mouth opening and masticatory muscle activity in cases of temporomandibular dysfunction (TMD) as compared to soft occlusive splints.

DETAILED DESCRIPTION:
A prospective, parallel randomized, controlled study will be conducted at the outpatient university clinic. Participant recruitment started following approval from the Ethics Committee .The patients will participate in the study after signing an informed consent form prior to data collection. Per inclusion criteria, subjects included are females less than 30 years of age, diagnosed with unilateral arthrogenous TMD, having complete permanent dentition and showing normal occlusion. Prior to participating in any study-related procedures, participants read and signed the informed consent form approved by the Institutional Review Board. Participants will be divided into three groups; three groups: LLLT (Group A); soft occlusive splint therapy OST (Group B); waitlist as controls (Group C).

Outcome measures: TMJ opening index (TOI), VAS, sEMG. Participants were not given information on which treatment they were receiving; they were only told that they could receive one of two different treatment techniques. Sessions were scheduled 3 days a week (every other day) for a total of 10 sessions

ELIGIBILITY:
Inclusion Criteria:

Females less than 30 years of age, Diagnosed with unilateral myogenous TMD, Having complete permanent dentition Showing normal occlusion

Exclusion Criteria:

Prior experience of Laser therapy, Systemic diseases (rheumatoid arthritis, ankylosing spondylitis, diabetes… etc. History of trauma in the TMJ or cervical regions; Neurological disorders, Muscular diseases; Cervical pain; Bruxism, Pregnancy; Currently on medication (analgesic, anti-inflammatory, muscle relaxants or anti- depressants) Current use of dental prosthetics; Previous orthodontal treatments; or Fixed restorations affecting occlusal surfaces.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Temporomandibular joint opening index (TOI): | baseline (pre-treatment) / after 3 weeks / and after 1 year
  Active and passive mouth opening will be assessed by a Boley gauge (Electronic Digital Caliper, CE Company, Japan)
  TOI= Passive opening mm -Maximum voluntary opening mm X 100 Passive opening mm +Maximum voluntary opening mm

SECONDARY OUTCOMES:
change in surface EMG (sEMG): | baseline (pre-treatment) / after 3 weeks / and after 1 year
  For recording, a surface electromyograph (Myotronics-Noromed, Inc., Tukwila WA, USA), with 8-channels, simultaneous acquisition, common grounding to all channels, and filters of 50 Hz electromyography with disposable electrodes will be used.
  Subjects will be seated on chairs with back and head rests to allow assessment from a relaxed position.
  The right masseter (RM), left masseter (LM), right anterior temporal (RAT), left anterior temporal (LAT), right sternocleidomastoid (RSM), and left sternocleidomastoid (LSM) muscles were recorded. The sEMG recordings and muscle activity will be expressed as the root mean square (rms) of the amplitude, expressed in µV.
Change in Visual Analogue Scale (VAS) | baseline (pre-treatment) / after 3 weeks / and after 1 year
  The pain VAS is a reliable measure of pain intensity with a 10 centimeters (100 mm) continuous scale attached by 2 verbal descriptors, one for each symptom extreme.
  For pain intensity, the scale is most anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100).
  The VAS only requires the ability to use a ruler to measure the distance to determine a score.

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Shousha, Principal Investigator — Lecturer
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
no plan to make individual participant data (IPD) available to other researchers